CLINICAL TRIAL: NCT04681898
Title: Incidence of Different Surgical Technics for Colorectal Deep Infiltrating EndoMetriosis on the Post-operative Fertility and Pregnancy Outcomes
Acronym: Endo-Metrios
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8088
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2020-11

CONDITIONS: Endometriosis
Keywords: colorectal endometriosis; deep infiltrating endometriosis; fertility; surgical technics in endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endometriosis is a disease that is very present on the current media scene. Its symptoms are very nonspecific and numerous. (dysmenorrhea, dyspareunia, dyschezia, urinary functional signs, infertility, chronic pelvic pain, etc.) Its prevalence is estimated at 10% of women and 20% of them have deep pelvic endometriosis. Colorectal lesions involving the rectosigmoid junction and the rectum represent the most severe forms and affect 5.3 to 12% of patients with deep pelvic endometriosis. Endometriosis is found in 20 to 50% of patients consulting for infertility and the rate of spontaneous pregnancy in patients with deep endometriosis is estimated to be between 8.7 and 13%. Surgery appears to improve fertility in women. However, several surgical techniques for deep endometriosis at the digestive level have been described, conservative or radical, without any having demonstrated its superiority both in terms of symptoms and fertility.

The aim of this study was to evaluate the incidence of different surgical technics (shaving vs. bowel resection) on post-operative fertility among patients with bowel deep infiltrating endometriosis and the pregnancy outcome

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (≥18 years old).
* woman with a desire to become pregnant and who had undergone surgery for the management of deep digestive endometriosis between September 01, 2009 and October 31, 2016.
* Woman who has not expressed, after information, the reuse of her data for the purposes of this research.

Exclusion Criteria:

* Woman who expressed her opposition to participating in the study
* Woman who had undergone a surgical intervention for the management of deep digestive endometriosis between September 01, 2009 and October 31, 2016 and having no desire to become pregnant
* Woman under safeguard of justice
* Woman under guardianship or guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult woman with a desire to become pregnant and who had undergone surgery for the management of deep digestive endometriosis between September 01, 2009 and October 31, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Retrospective analysis of the rate of occurrence of pregnancy postoperatively. | Files analysed retrospectily from September 1st, 2009 to October 31, 2016 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Émilie FALLER, Study Director — Department of Gynecology - Strasbourg University Hospitals
Locations (1):
- Department of Gynecology - Strasbourg University Hospitals, Strasbourg, France